CLINICAL TRIAL: NCT05185375
Title: Qualitative Analysis of Patients' Medical Records, to Understand the Reasons of the Difficulty in Controlling Asthma, in Difficult Forms
Brief Title: Qualitative Assessment of Patients Suffering From Difficult Asthma
Acronym: DIFFAsthme
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0727
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Asthma
Keywords: Severe, difficult-to-treat asthma; Difficult Asthma; Diagnosis; Comorbidities; Treatment; Allergy; Compliance
MeSH Terms: conditions — Asthma; Disease; Hypersensitivity; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is a chronic inflammatory disease, resulting from environmental, genetic and immunological factors. This is a triad specific to the diseases of the 21st century, linked to our environment, which the investigators thought were perfectly characterized and stable and which presents us with new challenges in their management. Our environment has not stopped changing over the past 30 years, so has our way of life and our way of working. The early detection of asthma and the initiation of an adequate therapy are most often carried out by primary care physicians, such as the general practitioner and the general pediatrician. These practitioners find themselves confronted with the medical complexity of asthma which essentially resides in the management of severe forms of asthma, defined by the high therapeutic charge needed to obtain a good control of the disease and, sometimes, in the management of difficult asthma which is an uncontrolled asthma independently of the patients' compliance and of the prescribed therapies. While general practitioners refer many cases of asthma to hospital experts, the investigators wanted to address the issue of difficult asthma, the management of which is less codified.

The main objective of this work is to identify, by a qualitative analysis of medical records, the profiles of patients referred for difficult asthma in a tertiary hospital in order, secondly, to target individual characteristics or subgroups on which therapeutic actions could be implemented, and to provide educational support for doctors.

ELIGIBILITY:
Inclusion criteria:

* Patients assessed for difficult asthma, from December 2015 to November 2020, at the University Hospital of Montpellier
* Patients aged from 5 to 99 years

Exclusion criteria:

* Patients not affiliated to French Social Security
* Patients not capable of understanding French
* Patients who don't have a diagnosis of difficult asthma

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting in the Respiratory Diseases outpatients Unit of the Arnaud de Villeneuve Hospital with a diagnosis of difficult-to-treat asthma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis of the medical records | day 1
  Qualitative analysis of the medical records from patients addressed to a tertiary hospital for difficult asthma

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC